CLINICAL TRIAL: NCT01141907
Title: Nurse-Led Heart Failure Care Transition Intervention for African Americans
Brief Title: Nurse-Led Heart Failure Care Transition Intervention for African Americans: The Navigator Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R21NR011056 (NIH); R21NR011056 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-06-11 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: heart failure; self care; decision support; telemonitoring; navigator
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Failure Self Care Support (Experimental): The goal of the Heart Failure Self Care Support Intervention (Navigator Program), delivered by a nurse and community health navigator team over 3 months post discharge from the index hospitalization, was to improve care transitions by providing patients with tools and support that promote knowledge and skills for HF self care as they transition from hospital to home. The multifaceted Navigator Intervention included the following intervention components: HF home automated telemonitoring support, medication and symptom self management, patient-centered record, HF care follow up, and activation of key supporter.
  Interventions: Behavioral: Heart Failure Self Care Support
- Usual Heart Failure Care (Active Comparator): Usual care for HF patients included the following: 1) Referral to HF clinic if the patient has no usual source of HF outpatient care, 2) HF patient education by HF care coordinator (advanced practice nurse), and 3) HF self care guide. All participants were treated by their usual source of HF care in the usual manner.
  Interventions: Other: Usual heart failure care

INTERVENTIONS:
Behavioral: Heart Failure Self Care Support — The intervention is aimed at preventing HF exacerbations and hospitalizations by improving self management with the support of the Home Automated Telemonitoring (HAT) system. The intervention was delivered by a RN-community health navigator (CHN) team over three months to HF patients and their caregivers in their home and via telephone and HAT system. The intervention was initiated during the index hospitalization. The RN-CHN team collaborated with participants, caregivers, and their usual source of HF care. Intervention strategies included tracking of weight and HF symptoms to provide feedback regarding self management and plan of care, enhancing medication and symptom self management, promoting HF care follow up, and promoting communication with providers.
  Arms: Heart Failure Self Care Support
Other: Usual heart failure care — Participants assigned to usual care are treated by their usual source of HF care in the usual manner and in accordance with the American College of Cardiology/American Heart Association Guidelines for the management of HF. Usual care for HF patients admitted to Johns Hopkins Hospital also includes the following: 1) Referral to HF clinic if the patient has no usual source of care and 2) HF patient education booklet.
  Arms: Usual Heart Failure Care

SUMMARY:
Heart failure (HF) affects over 5 million Americans with HF morbidity reaching epidemic proportions. Annual rates of new and recurrent HF events including hospitalization and mortality are higher among African Americans. In this study, the investigators are testing an interdisciplinary model for heart failure care, with focus on enhancing self management and use of telehealth, which has significant potential to improve self management and outcomes.

The main purpose of this study is to learn how to help African Americans with heart failure care for themselves at home. We hope to find out if a team including a nurse and community health navigator using a computer telehealth device can help people with heart failure stay healthier. The team will help people with heart failure to manage their medication, monitor their symptoms and weigh themselves every day after they leave the hospital. The team will also help people with heart failure learn to solve problems that may keep them from following their treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized with admitting diagnosis of heart failure in prior 8 weeks
* self-identified as African American
* community-dwelling (i.e., not in a long-term care facility)
* residence within a predefined radius in Baltimore City
* working telephone in their home
* provide signed informed consent

Exclusion Criteria:

* cannot speak or understand English
* severe renal insufficiency requiring dialysis
* acute myocardial infarction within preceding 30 days
* receiving home care services for HF post discharge
* legally blind or have major hearing loss
* screen positive for cognitive impairment on the Mini-cog at baseline
* unable to stand independently on a weight scale (limited ability to participate in HAT system)
* weigh more than 325 pounds (exceed scale capacity)
* serious or terminal condition such as psychosis or cancer (actively receiving chemo or radiation)
* pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl R Dennison, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Heart Failure Self Care Support: Navigator Team Intervention: The intervention is aimed at controlling heart failure (HF) and preventing exacerbations and hospitalizations by improving self management behaviors with the support of the Home Automated Telemonitoring (HAT) system. The intervention will be delivered by a RN-community health navigator (CHN) team over three months to HF patients and their caregivers in their home and via telephone and HAT system. The intervention will be initiated during the index hospitalization or as soon as possible after randomization. The RN-CHN team will collaborate with the participants, their caregivers, and their usual source of HF care. Intervention strategies include tracking of weight and HF symptoms to provide automated feedback regarding self management and plan of care, enhancing medication and symptom self management, promoting HF care follow up, and using a patient centered record to promote communication with providers.
Period: Overall Study
Arm/Group | Heart Failure Self Care Support | Usual Heart Failure Care
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heart Failure Self Care Support | Usual Heart Failure Care | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.4) | 56.8 (18.83) | 60.55 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rehospitalization
Description: Rehospitalization with primary diagnosis of heart failure
Time Frame: 3 months post enrollment
Measure: Number; unit: hospital readmisions
Arm/Group | Heart Failure Self Care Support | Usual Heart Failure Care
Number analyzed (Participants) | 6 | 5
hospital readmisions | 2 | 6

ADVERSE EVENTS:
Arm/Group | Heart Failure Self Care Support | Usual Heart Failure Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No